CLINICAL TRIAL: NCT06530251
Title: A Phase Ib/II Study of AK112 in Combination Therapy for Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Study of AK112 in Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-209
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AK112 in combination with AK130 (Experimental)
  Interventions: Drug: AK112; Drug: AK130
- AK112 in combination with AK127 (Experimental)
  Interventions: Drug: AK112; Drug: AK127
- AK112 in combination with Cadonilimab (Experimental)
  Interventions: Drug: AK112; Drug: Cadonilimab
- AK112 (Experimental)
  Interventions: Drug: AK112
- Sintilimab in combination with Bevacizumab biosimilar (Active Comparator)
  Interventions: Drug: Sintilimab Injection; Drug: Bevacizumab biosimilar

INTERVENTIONS:
Drug: AK112 — Following a predefined dose and date.
  Arms: AK112; AK112 in combination with AK127; AK112 in combination with AK130; AK112 in combination with Cadonilimab
Drug: Cadonilimab — Following a predefined dose and date.
  Arms: AK112 in combination with Cadonilimab
Drug: AK127 — Following a predefined dose and date.
  Arms: AK112 in combination with AK127
Drug: AK130 — Following a predefined dose and date.
  Arms: AK112 in combination with AK130
Drug: Sintilimab Injection — Following the local label direction.
  Arms: Sintilimab in combination with Bevacizumab biosimilar
Drug: Bevacizumab biosimilar — Following the local label direction.
  Arms: Sintilimab in combination with Bevacizumab biosimilar

SUMMARY:
There're 2 parts in this interventional study:

1. The goal of phase Ib trial is to evaluate the safety and tolerability of AK112 in combination therapies for the purpose of observing the incidence of dose limit toxicity (DLT) as well as the confirmation of maximum tolerable dose (MTD) in the treatment of advanced hepatocellular carcinoma (HCC), so as to determine the recommended phase 2 dose (RP2D) in the second part of the trial.
2. The goal of phase II trial is to evaluate the safety and efficacy of AK112 in combination therapy or monotherapy in the treatment of HCC compared to the combination of Sintilimab and Bevacizumab biosimilar.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent.
2. Have a life expectancy of at least 3 months.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. HCC confirmed by histology/cytology or confirmed by the American Society for the Study of Hepatology (AASLD) clinical diagnostic criteria for hepatocellular carcinoma in patients with cirrhosis.
5. Phase Ib:

   1. Barcelona Clinical Liver Cancer (BCLC) stage B or C.
   2. Has failed standard treatment and has received no more than two lines of anti-tumor treatment in the past;

   Phase II:
   1. The BCLC staging is stage C, which is not suitable for curative and local treatment, or for stage B that cannot be cured after curative and/or local treatment.
   2. Subjects who have not received any systematic anti-tumor treatment for HCC in the past.
6. According to RECIST v1.1, there is at least one untreatable measurable lesion, or a measurable lesion with clear imaging progression after local treatment, suitable for repeated and accurate measurement.
7. Liver function grading Child Pugh Grade A.
8. Has adequate organ function.
9. All subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.
10. Able to to comply with all requirements of study participation (including all study procedures).

Exclusion Criteria:

1. Components confirmed by histology/cytology, such as fibrous layer hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma.
2. Except for HCC, the subjects had other malignant tumors within the 5 years prior to enrollment. Subjects with other malignant tumors that have been cured through local treatment are not excluded, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast cancer in situ. If diagnosed with liver cancer or other malignant tumors more than 5 years before administration, pathological or cytological diagnosis of recurrent and metastatic lesions is required.
3. Tumor volume>50% liver volume; Portal vein cancer thrombus (Vp4), inferior vena cava cancer thrombus.
4. Tumors invade important organs and blood vessels around them, and researchers have determined that entering the study will cause a higher risk of bleeding.
5. There is central nervous system (CNS) metastasis, spinal cord compression, or meningeal metastasis.
6. There are pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage.
7. Previously received immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy, and any other treatments targeting the immune mechanisms of tumors.
8. Received local treatment for the liver within 4 weeks prior to the first administration; Received palliative radiotherapy for non liver patients within 2 weeks prior to initial administration.
9. There is a history of non infectious pneumonia that requires systemic glucocorticoid treatment, or current lung diseases including but not limited to interstitial lung disease, pneumoconiosis, silicosis, drug-related pneumonia, and severely impaired lung function.
10. History of severe bleeding tendency or coagulation dysfunction.
11. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia.
12. Any arterial or venous thromboembolism events, transient ischemic attacks, cerebrovascular accidents, hypertensive crises, or hypertensive encephalopathy occurred within 6 months prior to the first administration of medication.
13. Pregnant or lactating female subject.
14. Any prior or concurrent disease, treatment, or laboratory test abnormality that may confuse study results, affect subjects' full participation in the study, or may not be in their best interest to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | During the first three weeks.
  DLTs will be assessed during the first three weeks of treatment. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug.
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
Objective Response Rate (ORR) (Phase II) | Up to approximately 2 years.
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on RECIST Version 1.1).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Phase Ib) | Up to approximately 2 years.
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on RECIST Version 1.1).
Objective Response Rate (ORR) Per mRECIST | Up to approximately 2 years.
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on mRECIST).
Disease control rate (DCR) | Up to approximately 2 years.
  DCR is defined as the proportion of subjects with response of CR, PR and SD (based on RECIST Version 1.1).
Duration of Response (DoR) | Up to approximately 2 years.
  The time from first documented evidence of CR or PR until time of first documented disease progression.
Progression Free Survival (PFS) | Up to approximately 2 years.
  PFS is defined as the interval between first dose and the earliest date of disease progression or death due to any cause.
Time to response (TTR) | Up to approximately 2 years
  Time between date of start of treatment until first documented response (CR or PR).
Overall survival (OS) | From baseline until death due to any cause.
  OS is defined as the time from first dose until death due to any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute,Shandong Cancer Hospital), Jinan, Shandong